CLINICAL TRIAL: NCT05740696
Title: Registry Study for Optimal Management of Liver Failure in the Chinese Population (RESOLVE-C)
Brief Title: Registry Study for Optimal Management of Liver Failure in the Chinese Population
Acronym: RESOLVE-C
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-019
Record Dates: First submitted 2023-02-08; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-01

CONDITIONS: Liver Failure
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ALF: acute liver failure
  Interventions: Procedure: ALF
- SALF: subacute liver failure
  Interventions: Procedure: SALF
- ACLF: acute-on-chronic liver failure
  Interventions: Procedure: ACLF

INTERVENTIONS:
Procedure: ALF — Acute onset, no history of underlying liver disease, liver failure characterized by degree Ⅱ or above hepatic encephalopathy developed within 2 weeks
  Groups: ALF
Procedure: SALF — The onset was acute, with no history of underlying liver disease, and clinical manifestations of liver failure appeared between 2 and 26 weeks
  Groups: SALF
Procedure: ACLF — On the basis of chronic liver disease, the clinical manifestations of acute liver decompensation and liver failure appear in a short period
  Groups: ACLF

SUMMARY:
Liver failure is the most severe form of liver damage caused by viral, alcoholic, drug-related and ischemia-reperfusion factors, often combined with extrahepatic organ damage, resulting in a high mortality rate. This study intends to construct a real-world case registry database of inpatients with liver failure based on an electronic clinical data collection system through a multicenter collaborative network to study the clinical characteristics, epidemiology of bacterial and fungal infections, the impact of sarcopenia on clinical prognosis, and optimization of treatment strategies such as antiviral and artificial liver in Chinese inpatients with liver failure. The cohort and experience generated from this study will be used as a support for a series of future studies to focus on clinical issues such as infection, end-stage liver disease combined with organ failure, and early warning of critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

Patients with a diagnosis consistent with liver failure and pre-liver failure:

* Extreme weakness with significant gastrointestinal symptoms such as anorexia, vomiting and abdominal distention;
* Elevated alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) with progressive jaundice (TBil≥85.5 μmol/L);
* Bleeding tendency with PTA ≤ 60% or INR ≥ 1.5.

Exclusion Criteria:

* An event or complication that, in the judgment of the investigator, significantly affects the assessment of clinical status.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receive guideline-based systemic therapy. The follow-up assessments will be performed at week 1, 2, 3, 4, 12, 24 and 48 or any time if there is a change in condition. All the patients receive routine biochemical tests and imaging examinations.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 28-day
  28-day survival rates without liver transplantation
Overall survival | 90-day
  90-day survival rates without liver transplantation

SECONDARY OUTCOMES:
Disease progression | 48 weeks after discharge
  Incidence of complications and re-hospitalization at 48 weeks after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Yingli He, Pro., Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (14):
- China (14):
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Ankang Central Hospital, Ankang
  - Xiangya Hospital of Central South University, Changsha
  - Hanzhong 3201 Hospital, Hanzhong
  - Qilu Hospital of Shandong University, Jinan
  - First Hospital of Lanzhou University, Lanzhou
  - Weinan Central Hospital, Weinan
  - Air Force Medical University Tangdu Hospital, Xi'an
  - Shaanxi provincial people's hospital, Xi'an
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Xi 'an International Medical Center Hospital, Xi'an
  - Xianyang Central Hospital, Xianyang
  - The Affiliated Hospital of Yan'an University, Yanan
  - General Hospital of Ningxia Medical University, Yinchuan

REFERENCES:
- [Derived] Liu Y, Zhang Q, Li J, Wu X, Zang Q, Wang Q, Huang P, Wang Y, Zhang S, Liu S, Zhu C, Zhao Y, Yan T, He Y. mNGS improves the efficiency of infection diagnosis and treatment in acute-on-chronic liver failure. BMC Gastroenterol. 2026 Jan 20. doi: 10.1186/s12876-025-04601-8. Online ahead of print. PMID 41559596